CLINICAL TRIAL: NCT03878550
Title: Case-Control Study of the Glycotest™ HCC Panel Vs AFP for the Detection of Early-stage Hepatocellular Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Glycotest, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: G-1001
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Hepatocellular; Cirrhosis, Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Male and female adult patients with early-stage hepatocellular carcinoma against a background of liver cirrhosis.
- Controls: Male and female adult patients with liver cirrhosis at risk for hepatocellular carcinoma.

SUMMARY:
Clinical guidelines (AASLD) recommend the use of abdominal ultrasound (US) for surveillance testing for the early detection of Hepatocellular Carcinoma (HCC). The serum protein biomarker alpha-fetoprotein (AFP) is commonly used to augment US but its use alone is not recommended by clinical guidelines. Despite evidence that HCC surveillance improves early detection and reduces mortality from HCC, current HCC surveillance tests lack sensitivity, leaving a significant proportion of patients to present with late-stage disease. The Glycotest HCC Panel has shown better sensitivity than AFP, which is ineffective for the detection of early-stage HCC. This clinical study seeks to validate the Glycotest HCC Panel using a large multicenter cohort of cases and controls that includes patients diagnosed with early-stage HCC against a background of cirrhosis and cirrhotic patients without HCC (at risk) undergoing an established surveillance protocol.

DETAILED DESCRIPTION:
Study Rationale:

This study is designed to compare the ability of the Glycotest HCC Panel with that of AFP to differentiate between patients with early-stage Hepatocellular Carcinoma (HCC) against a background of cirrhosis from cirrhotic patients without HCC (at risk).

Primary Objective:

The primary objective of this study is to determine whether the Glycotest HCC Panel outperforms AFP in terms of area under the receiver operating characteristic curve (AUROC) for the differentiation of patients with early-stage HCC from those without HCC in the at-risk population.

Secondary Objective:

The secondary objective of this study is to determine whether the Glycotest HCC Panel outperforms AFP in terms of clinical sensitivity (as estimated using the 90% specificity estimate as the decision threshold) for the detection of patients with early-stage HCC.

Study Design:

This is a phase 2, multicenter, laboratory-blinded, case-control study of the Glycotest HCC Panel vs AFP for the discrimination of patients with early-stage HCC from those at risk. Case and control samples will be obtained from multiple institutions using prospective collection. The study will consist of a screening/baseline visit for all patients; controls initially assessed by abdominal US will also undergo a 6-month follow-up visit to confirm absence of HCC at enrollment. Assays will be performed by Glycotest with analysts blinded to clinical data.

Population:

The study population will comprise male and female adult patients with early-stage HCC against a background of cirrhosis (cases) as well as at-risk cirrhotic patients (controls). Enrollment of the aggregate of HCC cases with single lesions ≥ 3 cm and with multiple lesions will be capped at 50% of total cases. Enrollment of Chronic Hepatitis C cases and controls with sustained virologic response (SVR) to therapy will be matched. Cases and controls will be matched based on age, sex and etiology.

Number of Subjects:

Maximum of 388 cases and 378 controls;

* 150 cases and 140 controls (training set)
* Maximum of 238 cases and 238 controls (validation set)

Study Duration:

30 months ( approximately 24 months accrual + 6 month follow up)

Study Phases Patients potentially eligible for the study population will undergo informed consent prior to screening/baseline visits.

Screening Once consented, a subject's demographics, medical record, laboratory data, and imaging will be reviewed. Patients are considered eligible for enrollment once they meet all study enrollment criteria.

Enrollment Screening data will be re-reviewed if necessary and recorded. Serum from blood samples (5 mL) will be obtained for measurement of Glycotest HCC Panel score (which includes AFP).

Follow up Medical record review/imaging at 6 months from enrollment for control patients originally assessed using abdominal US.

ELIGIBILITY:
Inclusion Criteria:

Cases

1. Males and females ages 18 years or older.
2. Treatment-naïve HCC as defined by LI-RADS (Liver Imaging Reporting and Data System) LR-5 or OPTN (Organ Procurement and Transplantation Network) 5 CT or MRI criteria (all lesions must exhibit arterial phase hyper-enhancement), or histologic evidence.
3. Early-stage HCC defined by single lesion ≤ 5 cm or ≤ 3 lesions ≤ 3 cm determined at enrollment or within 100 days prior without vascular invasion.
4. Cirrhosis based on serum biomarkers (FibroSure®/FibroTest > 0.74, APRI (AST to Platelet Ratio Index) > 2, or FIB-4 (Fibrosis-4) > 3.25), histology, imaging, elastography, or clinical evidence of portal hypertension in the setting of known chronic liver disease.
5. Child-Pugh score A-B8.
6. Subject must be able to understand and provide informed consent.

Controls

1. Males and females ages 18 or older.
2. Cirrhosis based on serum biomarkers (FibroSure®/FibroTest > 0.74, APRI > 2, or FIB-4 > 3.25), histology, imaging, elastography, or clinical evidence of portal hypertension in the setting of known chronic liver disease.
3. Evidence of the absence of a solid hepatic mass, suspicious for HCC, at enrollment or within 100 days prior based on one of the following:

   1. Negative multiphase CT scan or MRI with contrast at screening/baseline visit, OR
   2. Negative abdominal US at both screening/baseline visit AND 6-month follow-up visit, OR
   3. Negative abdominal US at screening/baseline visit AND negative multiphase CT scan or MRI with contrast at 6-month or earlier follow-up visit.
4. Child-Pugh score A-B8.
5. Subject must be able to understand and provide informed consent.

Exclusion Criteria:

Cases

1. Uncontrolled ascites.
2. Uncontrolled encephalopathy.
3. History of liver transplant.
4. Diagnosis of active malignancy or history of active malignancy within 5 years prior to enrollment, including mixed HCC-CCA (cholangiocarcinoma). If previously diagnosed with malignancy, subject must be in remission for at least 5 years prior to enrollment. Prior history of HCC, including resection of HCC at any time, is excluded.
5. Prior treatment of tumor.
6. Any significant non-liver-related medical condition in which expected survival is less than 1 year.

Controls

1. Imaging evidence of solid hepatic mass, suspicious for HCC, including lesions meeting LI-RADS LR-3 or LR-4, OPTN-3 or OPTN-4, or LI-RADS LR-M criteria.
2. Uncontrolled ascites.
3. History of liver transplantation.
4. Uncontrolled encephalopathy.
5. Diagnosis of active malignancy or history of active malignancy within 5 years prior to enrollment (if previously diagnosed with malignancy, subject must be in remission for at least 5 years prior to enrollment). History of HCC including resection of HCC at any time, is excluded.
6. Any significant non-liver-related medical condition in which expected survival is less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise male and female adult patients with early-stage HCC against a background of cirrhosis (cases) as well as at-risk cirrhotic patients (controls). Enrollment of the aggregate of HCC cases with single lesions ≥ 3 cm and with multiple lesions will be capped at 50% of total cases. Enrollment of Chronic Hepatitis C cases and controls with sustained virologic response (SVR) to therapy will be matched. Cases and controls will be matched based on age, sex and etiology.
Sampling Method: Non-Probability Sample
Enrollment: 766 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AUROC | At enrollment
  Area under the receiver operating characteristics curve

SECONDARY OUTCOMES:
Sensitivity | At enrollment
  Clinical sensitivity for the detection of early-stage hepatocellular carcinoma as estimated using the 90% specificity estimate as the decision threshold

CONTACTS AND LOCATIONS:
Overall Officials: Josep Llovet, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jorge Marrero, MD, Principal Investigator — University of Pennsylvania Medical Center; Amit Singal, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (20):
- United States (19):
  - Cedars- Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Kaiser Permanente Northern California, San Francisco, California
  - University of California- San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - University of Florida, Gainesville, Florida
  - Miami VA Healthcare System, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania (HUP), Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Hebrew University- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang M, Sanda M, Comunale MA, Herrera H, Swindell C, Kono Y, Singal AG, Marrero J, Block T, Goldman R, Mehta A. Changes in the Glycosylation of Kininogen and the Development of a Kininogen-Based Algorithm for the Early Detection of HCC. Cancer Epidemiol Biomarkers Prev. 2017 May;26(5):795-803. doi: 10.1158/1055-9965.EPI-16-0974. Epub 2017 Feb 21. PMID 28223431